CLINICAL TRIAL: NCT04261348
Title: Effects of an Antimicrobial Stewardship (AMS) Program, on the Prevalence of Multidrug-resistant Gram - Negative Pathogens, in an Area of High Consumption of Antibiotics and High Resistance Rates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Sipsas, Professor, Laikο General Hospital, Athens
Other Study IDs: 59199
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Antimicrobial Stewardship Program

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
1. To evaluate the long-term effect of the AMS program on the consumption of broad-spectrum antibiotics and on the consumption of antibiotics in general (sustainability of the efficacy of the program). More specifically, the investigators shall examine the consumption of protected antibiotics during the years 2019 - 2020 and they shall compare it with the consumption of antibiotics before the implementation of the AMS program.
2. To evaluate the impact of the AMS program, combined with an infection control program, on the incidence of MDRGN infections in a hospital with high MDR incidence. Confounding factors are a barrier to analyze the impact of ASPs on antibiotic resistance. In a hospital setting, one of the most important confounding factors is the implementation of infection control practices at the same time as the ASPs. It is extremely difficult to infer causality between an ASP and antibiotic resistance reduction when infection control is a confounding factor, especially if the study intervention combines an ASP and infection control practices performed at the same time. The way to go around the problem is to implement ASP and IC at different time points. The investigators implemented the ASP program in September 2015 and they added the IC program in September 2018. Therefore, the investigators shall be able to compare the two-time periods (i.e. ASP alone vs. ASP/IC) by using the time series analysis and delineate the impact of each intervention.
3. To evaluate the effect of the AMS program on patient outcomes (in-hospital mortality, length of stay)

ELIGIBILITY:
Inclusion Criteria:

NA

Exclusion Criteria:

NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will be administered antibiotics
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Consumption of antibiotics | 2 years
  consumption of antimicrobials (defined daily doses / 100 patient-days)
Days of therapy | 2 years
  days of therapy for each drug (number of days)
Days of antibiotics | 2 yars
  days of antibiotics (number of days)
Patients receiving surgical prophylaxis | 2 years
  percentage of patients receiving appropriate surgical prophylaxis
Hospital mortality rate | 2 years
  in-hospital mortality rate (%)
Clinical cure rate | 2 years
  clinical cure rate of the initial antibiotic regimen (%)
Length of stay | 2 years
  length of stay (number of days)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Laikon, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No